CLINICAL TRIAL: NCT03170258
Title: Self-activation of Reward-related Brain Regions in Individuals With and Without Nicotine Dependence
Brief Title: Self-activation in Individuals With and Without Nicotine Dependence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unanticipated difficulty with enrollment
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Brain & Behavior Research Foundation (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00081458; UL1TR001117 (NIH); 24393 (Other Grant/Funding Number: Brain & Behavior Research Foundation)
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Addiction Nicotine
Keywords: real-time fMRI; reward; motivation; dopamine; EEG
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Reward-related Brain Region Feedback (Experimental): Participants in this group will receive neurofeedback from a reward-related brain area (e.g., VTA, PFC) using EEG and/or fMRI during the experiment.
  Interventions: Device: Neurofeedback (from fMRI and/or EEG)
- Noise Control (Sham Comparator): Participants in this group will receive sham neurofeedback. Participants will be debriefed at the end of the study.
  Interventions: Device: Neurofeedback (from fMRI and/or EEG)

INTERVENTIONS:
Device: Neurofeedback (from fMRI and/or EEG) — During part of the task, a feedback display (e.g., thermometer stimulus) will be used to display the average brain activity for each participant. This signal will be acquired ~ every 1 second during the neurofeedback session and will dynamically update to reflect ongoing changes in brain activity. This continuously updated display is the primary feedback mechanism provided to the participant.

SUMMARY:
The purpose of this study is to see if a non-medication intervention can increase motivation and reward processing to non-drug reward cues (for example, a picture of one's favorite food) in individuals with and without nicotine dependence by observing brain activity using electroencephalography (EEG) and/or functional magnetic resonance imaging (fMRI). The investigators hypothesize that learning to increase brain activity to non-drug cues may improve reward responses and motivation to non-drug cues, and for individuals who smoke, may eventually result in improved smoking cessation outcomes.

DETAILED DESCRIPTION:
The purpose of this study is to:

1. Assess the ability of adults with and without nicotine dependence (ND) to activate reward-related brain regions (e.g., ventral tegmental area (VTA), striatum, prefrontal cortex).
2. Evaluate whether fMRI and/or EEG neurofeedback improves the ability to increase reward-related brain activation in individuals with and without ND.
3. Examine the relationship between activation of reward-related regions via neurofeedback and dopamine availability (as assessed genetically).
4. Examine the effects of neurofeedback on clinically relevant outcomes, including reward responsivity and smoking related behaviors.

Procedure:

Prior to coming to a screening visit, all potential participants will undergo a phone pre-screening using an IRB approved phone script to pre-identify potentially eligible participants and to potentially decrease screen fail rate. These interested potential participants call or email the site in response to advertisements. The pre-screening will take place via phone. Participants who pass the pre-screening will complete some or all of the following visits: Screening, Camera Return Visit, Real-Time Neurofeedback Visit, Follow-up Phone Call/Debriefing.

Screening Visit:

Participants with nicotine dependence who pass the pre-screen will come to the lab at Duke to complete additional screening. All participants will undergo informed consent and those with ND will complete a urine drug screen. Participants who pass the urine drug screen (results are provided immediately) will complete questionnaires assessing mood, reward processing, and smoking behaviors.

Some participants may also be given a camera to use to capture pictures of personalized rewarding objects (e.g., picture of their pet, favorite book, favorite food). Participants may be loaned the camera for a period of 1-2 weeks to capture pictures of rewarding objects. We will instruct participants that the camera is to be used exclusively for capturing pictures for the study and not for personal use. Some participants may not be asked to take their own pictures for the study protocol and may simply be shown neutral or positive pictures/images/objects provided by the experimenters (e.g., shapes, pictures, etc.). Note, no aversive images will be shown to participants.

Camera Return Visit:

Participants who were loaned a camera will be asked to come to the lab at Duke to return the camera. The experimenters will ensure that enough pictures have been acquired to use during the experiment. Participants will be given guidelines about what types of pictures are required for the study. Participants are also free to provide photos they already have by uploading them to a secure website or brining them in on a device (e.g., thumbdrive).

Participants may also be asked to view and rate the pictures they provide along with neutral and positive images we provide (e.g., puppy, flower) on dimensions such as valence and arousal.

Real-Time Neurofeedback Visit:

Eligible participants will be scheduled for an fMRI and/or EEG session to assess and measure the ability to self-activate reward-related regions. The fMRI session will be conducted at the Duke Brain Imaging and Analysis Center (BIAC) and/or the UNC Biomedical Research Imaging Center (BRIC). Female participants will have a urine pregnancy test prior to fMRI scanning; the test will be verified to be negative in order to proceed with the scanning session. The EEG sessions will take place in private testing space in the Levine Science Research Center or the BIAC.

Participants may complete some or all of the following tasks: Reward Activation Task, Passive Viewing Task, and Reward Learning Task. All of these tasks aim to assess how adults can learn to interact with neurofeedback provided from an fMRI or EEG system. The tasks vary slightly from each other in terms of stimuli used (personalized pictures, images provided by the experimenters, feedback display, etc.). It may be possible that we will not be able to get a good EEG signal for some participants, based on equipment error or head size. If this occurs, participants will be debriefed. We will be sure to emphasize there was no error on the participant's part, and that sometime the signal is difficult to acquire for a variety of reasons.

ELIGIBILITY:
Inclusion Criteria:

1. 18-45 years of age
2. Right handed
3. In good general health
4. Male or Female
5. For ND individuals: Self-reported smoking ≥ 5 combustible cigarettes per day
6. For ND individuals: Afternoon expired CO concentration of ≥ 8 ppm
7. For ND individuals: Is willing and able to abstain from smoking for a few hours

Exclusion Criteria:

1. History of chronic/significant medical condition
2. Current or past 6 month use of prescription medications for psychiatric conditions (e.g., depression, anxiety)
3. Current or past 6 month diagnosis of anxiety, bipolar disorder, depression, OCD, schizophrenia, psychosis, or personality disorder.
4. Current substance abuse or dependence or history within the last 6 months (other than nicotine for ND individuals)
5. For ND individuals: Positive drug test for anything other than marijuana
6. For ND individuals: Currently on nicotine replacement therapy
7. For ND individuals: Individuals who role their own cigarettes
8. For ND individuals: Daily cannabis use
9. For ND individuals: Consume more than 21 alcoholic drinks per week
10. For ND individuals: Use harder drugs (e.g., cocaine, methamphetamine) more than 10 times per year
11. For ND individuals: Currently taking medication that directly acts on the dopamine system (e.g., L-DOPA).
12. Inability to understand written and/or spoken English language
13. For MRI subjects: Claustrophobia or other contraindications to MRI scanning
14. For MRI subjects: If female, pregnancy as determined by urine pregnancy test on the day of MRI scanning
15. For MRI subjects: Presence of any metal in the body (e.g., implant, non-removable piercing, metal IUD)
16. For MRI subjects: Head injury resulting in loss of consciousness
17. For MRI subjects: Worked with metal (e.g., welding) or had an injury to the eye involving metal
18. For MRI subjects: Weigh more than 250 pounds

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Alison Adcock, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Center for Cognitive Neuroscience, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to upload the fMRI statistical image maps on NeuroVault. We will do so after data collection is complete.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Duke University community and surrounding Durham area via flyers, print advertisements, online advertisements, and word of mouth. To qualify for the study, subjects who smoke must self-report smoking greater than or equal to 5 cigarettes per day and be in good health.
Pre-assignment Details: No participants were randomized to the Noise Control arm.
Period: Overall Study
Arm/Group | Reward-related Brain Region Feedback | Noise Control
Started | 46 | 0
Completed | 39 | 0
Not Completed | 7 | 0
Not completed — Physician Decision | 4 | 0
Not completed — Equipment issues | 1 | 0
Not completed — Medication | 1 | 0
Not completed — Sleep issues | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Reward-related Brain Region Feedback
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 16
  More than one race | 3
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Reward-related Brain Activation as Measured by fMRI
Description: The investigators will examine the change in brain activation in the target region (e.g., VTA) during the task. This includes prior to, during, and following real-time neurofeedback. Reported is the percent signal change from baseline (last 3 volumes of prior count condition).
Time Frame: Changes will be assessed across the task (~30 minutes) during the neurofeedback visit
Population: Of the total number of completed participants (n=39), 5 participants completed data collection for the fMRI portion.
Measure: Mean (Standard Deviation); unit: percentage of signal change
Arm/Group | Reward-related Brain Region Feedback
Number analyzed (Participants) | 5
percentage of signal change | 0.4864 (0.4798)
Statistical Analysis 1: Comparison: Reward-related Brain Region Feedback; Test type: Other; p = 0.0015, t-test, 2 sided; One-sample 2-sided t-test against a mean of 0 used to evaluate the main effect of VTA activation during neurofeedback

2. Primary Outcome: Change in Reward-related Brain Activation as Measured by EEG Ratio of Beta to Theta Power
Description: The investigators will examine the change in brain activation in the target region (e.g., VTA) during the task. This includes prior to, during, and following real-time neurofeedback. Reported here is the change from baseline (prior to real-time neurofeedback) and ~30 minutes following real-time neurofeedback. The ratio of Beta to Theta power indicates the level of active brainwave activity (Beta) versus the level of resting brainwave activity (Theta).
Time Frame: Baseline (prior to real-time neurofeedback) and ~30 minutes following real-time neurofeedback
Population: Of the total number of completed participants (n=39), 34 total participants completed data collection for the EEG portion; 6 participants included in analysis due to data quality.
Measure: Mean (Standard Deviation); unit: ratio of Beta to Theta power
Arm/Group | Reward-related Brain Region Feedback
Number analyzed (Participants) | 6
ratio of Beta to Theta power | 0.13 (0.12)
Statistical Analysis 1: Comparison: Reward-related Brain Region Feedback; Test type: Other; p > 0.10, t-test, 1 sided; One-sample t-test against 0 for the ratio of Beta to Theta power

3. Secondary Outcome: Dopamine Availability
Description: Dopamine availability as assessed by genetic saliva samples
Time Frame: Collected once during the screening visit
Population: Saliva samples not collected due to safety procedure during COVID-19 pandemic.
Arm/Group | Reward-related Brain Region Feedback
Number analyzed (Participants) | 0

4. Secondary Outcome: Onset to Smoking a Cigarette
Description: The time (in minutes) to when participants smoke their first cigarette following the MRI session
Time Frame: up to 30 minutes following the neurofeedback session
Population: Participants who chose to smoke a cigarette after the MRI session.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Reward-related Brain Region Feedback
Number analyzed (Participants) | 2
minutes | 1.00 (1.41)

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Arm/Group | Reward-related Brain Region Feedback
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/58/NCT03170258/Prot_SAP_000.pdf